CLINICAL TRIAL: NCT05504304
Title: Outcomes of Sanders Type IV Calcaneal Fractures Treated With Open Reduction and Internal Fixation (ORIF) Plus Primary Subtalar Arthrodesis (PSTA) Versus Conservative Management Then Calcaneoplasty and Late Subtalar Arthrodesis.
Brief Title: Primary Subtalar Arthrodesis Versus Late Subtalar Arthrodesis in Sanders Type IV Calcaneal Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Bishoy Emil, assistant lecturer, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD
Record Dates: First submitted 2022-07-31; First posted 2022-08-17 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Calcaneus Fracture
Keywords: Primary subtalar arthrodesis; Late subtalar fusion
MeSH Terms: interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: open reduction and internal fixation plus primary subtalar arthrodesis. (Active Comparator): they will be scheduled to surgery after resolution of the edema and appearance of wrinkle sign. Lateral position and lateral extensile approach will be used. A 4 mm schanz will be inserted in the calcaneal tuberosity from lateral side to control varus and to restore calcaneal height. Lateral wall of the calcaneus will be lifted keeping it attached inferiorly. Articular surfaces of inferior surface of the talus and posterior facet of the calcaneus will be debrided thoroughly and drilled by 2 mm k-wire. tricortical iliac bone autograft will be inserted the subtalar joint. A lateral nonlocked plate will be applied to reduce the lateral wall blow out and broadening then fixation by two cannulated partially threaded 7.3 screws from the calcaneal tuberosity to the talus. We will check position by fluoroscopy then closure in two layers (subcutaneous and skin) after homeostasis. Below knee slab will be applied and non-weight bearing for six weeks.
  Interventions: Procedure: open reduction and internal fixation plus primary subtalar arthrodesis
- Group B: conservative management then calcaneoplasty and subtalar arthrodesis. (Active Comparator): they will be assessed upon 1st clinic visit. After at least three months patients will be scheduled for subtalar arthrodesis. A new preoperative ankle CT scan will be done. Lateral position and lateral extensile approach will be used. Lateral wall and plantar exostosis will be resected. Articular surfaces of inferior surface of the talus and posterior facet of the calcaneus will be debrided thoroughly and drilled by 2 mm k-wire. Hind foot deformity (mostly varus) will be corrected through the subtalar joint manually and checked clinically. Loss of calcaneal height will be corrected by tricortical iliac bone autograft to distract the subtalar joint then fixation by two cannulated partially threaded 7.3 screws from the calcaneal tuberosity to the talus. We will check position by fluoroscopy then closure in two layers (subcutaneous and skin) after homeostasis. Below knee slab will be applied and non-weight bearing for six weeks.
  Interventions: Procedure: conservative management then calcaneoplasty and subtalar arthrodesis.

INTERVENTIONS:
Procedure: open reduction and internal fixation plus primary subtalar arthrodesis — they will be scheduled to surgery after resolution of the edema and appearance of wrinkle sign. Lateral position and lateral extensile approach will be used. A 4 mm schanz will be inserted in the calcaneal tuberosity from lateral side to control varus and to restore calcaneal height. Lateral wall of the calcaneus will be lifted keeping it attached inferiorly. Articular surfaces of inferior surface of the talus and posterior facet of the calcaneus will be debrided thoroughly and drilled by 2 mm k-wire. tricortical iliac bone autograft will be inserted the subtalar joint. A lateral nonlocked plate will be applied to reduce the lateral wall blow out and broadening then fixation by two cannulated partially threaded 7.3 screws from the calcaneal tuberosity to the talus. We will check position by fluoroscopy then closure in two layers (subcutaneous and skin) after homeostasis. Below knee slab will be applied and non-weight bearing for six weeks.
  Arms: Group A: open reduction and internal fixation plus primary subtalar arthrodesis.
Procedure: conservative management then calcaneoplasty and subtalar arthrodesis. — they will be assessed upon 1st clinic visit. After at least three months patients will be scheduled for subtalar arthrodesis. A new preoperative ankle CT scan will be done. Lateral position and lateral extensile approach will be used. Lateral wall and plantar exostosis will be resected. Articular surfaces of inferior surface of the talus and posterior facet of the calcaneus will be debrided thoroughly and drilled by 2 mm k-wire. Hind foot deformity (mostly varus) will be corrected through the subtalar joint manually and checked clinically. Loss of calcaneal height will be corrected by tricortical iliac bone autograft to distract the subtalar joint then fixation by two cannulated partially threaded 7.3 screws from the calcaneal tuberosity to the talus. We will check position by fluoroscopy then closure in two layers (subcutaneous and skin) after homeostasis. Below knee slab will be applied and non-weight bearing for six weeks.
  Arms: Group B: conservative management then calcaneoplasty and subtalar arthrodesis.

SUMMARY:
Fracture calcaneus accounts for up to 2% of all fractures. 75% of calcaneal fractures are displaced intra-articular fractures and historically have been associated with poor functional outcomes.

When the talus applies an axial loading to the posterior facet, shear forces result in a primary fracture line between medial (sustentaculum tali) and lateral part of the calcaneus. As the axial force continues, a secondary fracture line will develop. According to the relation of the secondary fracture line's exit to insertion of tendo-achilis Essex-Lopresti classified that into two types joint depression and tongue.

Numerous classifications exist in the literature but that by Sanders is the most prevalent and best suited for clinical practice and for research purposes.

Sanders in his clinical trials found that as the number of articular fragments- based on axial and coronal CT scan cuts with the widest undersurface of the posterior facet of the talus- increase, the results and prognosis worsen.

Up to 73% in the sanders type IV fractures eventually leads to subtalar fusion to manage post-traumatic subtalar arthritis. They are 5.5 times more likely to require subtalar arthrodesis than Sanders II fractures. Second surgeries increase the cost of management and delay the return of level of function for the patient.

Some authors advocate that the fractures with a higher Sanders classification demonstrated no difference between operative and non-operative treatment. However, careful stratification of the patients may show better outcomes after surgical intervention in some groups.

There is no consensus about how to manage calcaneal fractures but we can divide management into four broad categories: Non-operative, Open reduction and internal fixation, Minimally invasive reduction and fixation and finally Primary ORIF and subtalar arthrodesis.

Our trial was conducted to add to the current evidence and our main questions are: does initial reduction and fixation of comminuted displaced intra-articular Sanders type IV calcaneal fractures matter in subtalar fusion?

DETAILED DESCRIPTION:
Randomization: patients presented to clinic or emergency room with recent (30 days or less) Sanders type IV intra-articular calcaneal fractures will be included in group A. Patients referred to our clinic (from other surgeons or hospitals) with old (more than three months) Sanders type IV intra-articular calcaneal fractures will form group B.

Group A: open reduction and internal fixation plus primary subtalar arthrodesis.

Group B: conservative management for at least three months then calcaneoplasty and late subtalar arthrodesis.

Ethical Considerations: Will be followed by obtaining the hospital Research Ethics Committee approval and written informed consents from the patients.

Intervention:

All patients were subjected to the same initial treatment with below knee slab, limb elevation and analgesics.

Patient in group A will be scheduled to surgery after resolution of the edema and appearance of wrinkle sign.

They will be anesthetized and tourniquet will be applied over the thigh. Lateral position and lateral extensile approach will be used. A full flap will be developed by subperiosteal dissection with protection of sural nerve and peroneal tendons. Three k-wires will be inserted in fibula, lateral surface of talus and cuboid bones as retractors.

A 4 mm schanz will be inserted in the calcaneal tuberosity from lateral side to control varus and to restore calcaneal height. Lateral wall of the calcaneus will be lifted keeping it attached inferiorly. Articular surfaces of inferior surface of the talus and posterior facet of the calcaneus will be debrided thoroughly and drilled by 2 mm k-wire. tricortical iliac bone autograft will be inserted the subtalar joint. A lateral nonlocked plate will be applied to reduce the lateral wall blow out and broadening then fixation by two cannulated partially threaded 7.3 screws from the calcaneal tuberosity to the talus. We will check position by fluoroscopy then closure in two layers (subcutaneous and skin) after homeostasis. Below knee slab will be applied and non-weight bearing for six weeks.

Group B patients will be assessed upon 1st clinic visit. After at least three months patients will be scheduled for subtalar arthrodesis. A new preoperative ankle CT scan will be done.

Patients will be anesthetized and tourniquet will be applied over the thigh. Lateral position and lateral extensile approach will be used. A full flap will be developed by subperiosteal dissection with protection of sural nerve and peroneal tendons. Three k-wires will be inserted in fibula, lateral surface of talus and cuboid bones as retractors.

Lateral wall and plantar exostosis will be resected. Articular surfaces of inferior surface of the talus and posterior facet of the calcaneus will be debrided thoroughly and drilled by 2 mm k-wire. Hind foot deformity (mostly varus) will be corrected through the subtalar joint manually and checked clinically. Loss of calcaneal height will be corrected by tricortical iliac bone autograft to distract the subtalar joint then fixation by two cannulated partially threaded 7.3 screws from the calcaneal tuberosity to the talus. We will check position by fluoroscopy then closure in two layers (subcutaneous and skin) after homeostasis. Below knee slab will be applied and non-weight bearing for six weeks.

Post operatively, both groups will be followed after intervention every two weeks for two months then every three months for one year. Outcomes will be assessed using questionnaires in our clinic at six months and one-year visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a Sanders IV displaced intra-articular calcaneal fracture (DIACF).
* Within 12 months from injury.
* Clear demonstration of at least 3 fracture lines across the posterior subtalar facet, dividing it into at least 4 fragments and the fragments being displaced by at least 2 mm, as seen on the coronal and axial CT scans (classified as Sanders IV).
* Ability to provide informed consent.
* Available for follow-up for at least 6 months after intervention.

Exclusion Criteria:

* Medical contraindications to surgery.
* Fracture more than 12 months old at first presentation.
* Previous calcaneal pathology (infection, tumor etc).
* Previous calcaneal surgery.
* Co-existent foot or ipsilateral lower limb injury.
* Open calcaneal fractures.
* Inability to obtain preoperative CT scans or accurately classify the fractures as per Sanders classification system.

Ages: 16 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
the American Orthopaedic Foot and Ankle Society's Ankle-Hindfoot score (AOFAS score) | up to two years
  functional state of the patient
Foot and Ankle Ability Measure (FAAM). | up to two years
  functional state of the patient
time to return to work in months | up to two years
  the time from injury till resuming their jobs (if returned to job)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
if needed will be shared as excel sheets
Supporting Information: Study Protocol, SAP
Time Frame: after publication
Access Criteria: open access